CLINICAL TRIAL: NCT02944890
Title: A Multicenter, Randomized, Controlled Study to Compare the Efficacy and Safety of 2 Types of Drug Eluting Balloon Catheters (RESTORE DEB and SeQuent® Please) in Chinese Patient With Coronary In-stent Restenosis (ISR)
Brief Title: Compare the Efficacy and Safety of RESTORE DEB and SeQuent® Please in Chinese Patient With Coronary In-stent Restenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZhuHai Cardionovum Medical Device Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG01W-1101
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2017-07

CONDITIONS: Coronary Restenosis
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- RESTORE DEB (Experimental): Conduct Drug Eluting Balloon Catheters(RESTORE DEB）
  Interventions: Device: Drug Eluting Balloon Catheters(RESTORE DEB）
- SeQuent® Please (Active Comparator): Conduct Drug Eluting Balloon Catheters(SeQuent® Please）
  Interventions: Device: Drug Eluting Balloon Catheters(SeQuent® Please）

INTERVENTIONS:
Device: Drug Eluting Balloon Catheters(RESTORE DEB）
  Arms: RESTORE DEB
Device: Drug Eluting Balloon Catheters(SeQuent® Please）
  Arms: SeQuent® Please

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Paclitaxel drug eluting balloons (RESTORE DEB, 3μg/mm2 balloon surface area ) for success of intervention treatment and maintaining the vessels unobstructed in the treatment of coronary in-stent restenosis compared with a product of the same category (SeQuent® Please).

ELIGIBILITY:
Inclusion Criteria:

Related to the patients:

1. Age ≥18 years old
2. Patients agree to receive follow-ups in month-1, 6, 9 and 12, and receive angiography in month-9.
3. Patients are able to understand the objectives of the study mentally and in language. Patients should indicate sufficient compliance to the study, and acknowledge all risks and benefits by signing the informed consent form.
4. Patients with stable angina pectoris, or unstable angina pectoris, or old myocardial infarction, or proved asymptomatic regional myocardial ischemia
5. Patients suitable to receive coronary revascularization of any type (including balloon angioplasty, stent implantation or coronary artery bypass grafting)

   Related to the diseases:
6. Restenosis Mehran type I-III after stent implantation (including bare metal stents, stents with inert coating, and stents with active coating) for the first time
7. Diameter of the stent with restenosis should be 2.5-4.0mm (included). Length of the stenosis lesion should be no more than 26mm, and diameter stenosis before operation should be ≥70%, or ≥50% with the evidence of ischemia.
8. One subject is allowed to have 2 target lesions at most, and 2 Paclitaxel drug balloons for dilation.
9. The distance between lesions which require intervention and the target lesions must be >10mm.

Exclusion Criteria:

Related to the patients:

1. Pregnant or lactating women, or women who plan to get pregnant within 12 months or refuse to take effective contraceptives.
2. The patients are participating in any other clinical trials before reaching the primary endpoints.
3. The patients have a life expectancy of less than 12 months, or it would be difficult to finish follow-ups within 12 months.
4. The patients had cerebral stroke within 6 months before being included, or have a history of peptic ulcer or gastrointestinal bleeding in the past 6 months, or the patients have a bleeding tendency according to the investigator.
5. Patients with a history of leukopenia (white blood cell count <3×109/L for more than 3 days) or neutropenia (ANC<1000/mm3 for more than 3 days) or thrombocytopenia (platelet <100,000/mm3)
6. Patients who are forbidden to use anticoagulation agents or anti-platelet drugs, and unable to tolerate Aspirin or Clopidogrel
7. Patients with renal insufficiency (eGFR<30mL/min)
8. Patients who are known to be allergic to Paclitaxel
9. Patients who had myocardial infarction within 1 week before being included
10. Patients who had heart transplantation
11. Patients with severe congestive heart failure or NYHA grade IV heart failure
12. Patients with severe valvular heart disease
13. Patients who are unsuitable for the study according to the investigator due to other reasons

    Related to the diseases:
14. Patients with evidence of extensive thrombosis in the target vessel before intervention
15. Patients with total occlusion indicating TIMI 0 blood flow at the target lesion (Mehran type IV stenosis)
16. Patients with multiple lesions (≥3) requiring percutaneous coronary intervention treatment in the same artery
17. Patients with lesions requiring intervention treatment in 3 vessels
18. The diameter of the branch lesions in the target lesion ≥2.5mm
19. Patients already treated with CABG after in-stent restenosis
20. LM lesions and Ostial lesion within 5mm to the root aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss of the target lesion | 9 months

SECONDARY OUTCOMES:
The success rate of intervention treatment: including device success, lesion success and clinical success | 1-2 days
Occurrence rate of restenosis in the target lesions | 9 months after the operation
Target lesion revascularization (TLR) rate | 1, 6, 9, and 12 months after the operation
Target vessel revascularization (TVR) rate | 1, 6, 9, and 12 months after the operation
Target lesion failure (TLF) rate | 1, 6, 9, and 12 months after the operation
Occurrence rate of major adverse cardiovascular events | 1, 6, 9, and 12 months after the operation
All adverse events and severe adverse events | 1, 6, 9, and 12 months after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (14):
- China (14):
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Tangdu Hospital, Xi'an, Shaanxi
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital School of medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Chen Y, Gao L, Qin Q, Chen S, Zhang J, Chen H, Wang L, Jin Z, Zheng Y, Zhang Z, Li H, Li X, Fu G, Chen L, Sun Z, Wang Y, Jin Q, Cao F, Guo J, Zhao Y, Guan C, Li W, Xu B; RESTORE ISR China Investigators. Comparison of 2 Different Drug-Coated Balloons in In-Stent Restenosis: The RESTORE ISR China Randomized Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2368-2377. doi: 10.1016/j.jcin.2018.09.010. PMID 30522665